CLINICAL TRIAL: NCT02830425
Title: Potentially Inappropriate Prescription Associated to Multimorbidity, Using the Explicit STOPP-START (Screening Tool of Older Persons' Potentially Inappropriate Prescriptions/Screening Tool to Alert Doctors to the Right Treatment) Criteria
Brief Title: Potentially Inappropriate Prescription Associated to Multimorbidity
Acronym: PIMyC
Status: Completed | Type: Observational
Sponsor: Corporacion Parc Tauli (Other)
Collaborators: Fondo de Investigacion Sanitaria (Other); Hospital del Mar (Other); Hospital de Galdakao (Other); Consorci Hospitalari de Vic (Other); Hospital Universitario de Canarias (Other)
Responsible Party: Principal Investigator, Marisa Baré, MD, MPH, PhD, Cancer Screening-Epidemiology Coordinator, Corporacion Parc Tauli
Other Study IDs: PI15/00552
Record Dates: First submitted 2016-07-01; First posted 2016-07-12 (Estimated); Last update posted 2020-04-09 (Actual); Status verified 2020-04

CONDITIONS: Chronic Disease
Keywords: Multimorbidity; Polypharmacy; Appropriateness; STOPP; START
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Other: No intervention

SUMMARY:
A prospective multicenter cohort study in 5 hospitals in Spain will be initiated in 2016.

Objectives:

1. To estimate and describe patterns of multimorbidity and polypharmacy in patients over 64 admitted for a chronic disease exacerbation.
2. To analyze the potentially inappropriate prescribing (PPI) drugs according to STOPP / START (SS) criteria.
3. To evaluate the relationship between multimorbidity and PPI and adverse medication (RAM) preventable reaction.

The cohort will include 800 patients >64 years admitted in internal medicine and / or geriatric department of 5 hospitals of the National Health Service. Application of the SS criteria (released in 2015) on admission and at discharge, and collection of demographic and clinical variables including comorbidities, baseline chronic medication, geriatric syndromes, functional capacity and RAM. Descriptive analysis and bivariate parametric or nonparametric tests will be applied to analyze relationship between morbidity, polypharmacy, SS criteria and RAM. Intraobserver agreement will be assessed for SS criteria. Multiple regression techniques will be applied, where the dependent variable will be the PPI or the RAM.

ELIGIBILITY:
Inclusion Criteria:

* Patient admitted to the Internal Medicine or Geriatrics department
* Admitted to hospital because of an exacerbation of any previous chronic condition

Exclusion Criteria:

* Terminal ill patients at admission
* Patients with lower forecast life than 1 year
* Patient admitted to the hospital only because an acute problem
* In patient home care

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Elderly with any chronic condition admitted in Internal Medicine or Geriatrics department because of an exacerbation of any chronic condition
Sampling Method: Non-Probability Sample
Enrollment: 740 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2019-07 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with Potentially inappropriate medication, according to STOPP-START explicit criteria | At study entry

SECONDARY OUTCOMES:
Percentage of patients with Potentially inappropriate medication, according to STOPP-START explicit criteria | Through study completion, an average of 2 years
Percentage of patients with polypharmacy | At study entry
  Polypharmacy=more than 5 chronic medications
Patients with any treatment-related adverse events (ADR), according to the Wills & Brown classification | Through study completion, an average of 2 years
Percentage of different Patterns of multimorbidity in chronic patients, according to clusters or associations of different chronic conditions | At study entry

CONTACTS AND LOCATIONS:
Overall Officials: Marisa Baré, MD, MPH, PhD, Principal Investigator — Corporacio Parc Taulí
Locations (1):
- Corporacio Parc Taulí, Sabadell, Spain

REFERENCES:
- [Background] Bare M, Herranz S, Jordana R, Gorgas MQ, Ortonobes S, Sevilla D, De Jaime E, Ibarra O, Martin C; MoPIM study group. Multimorbidity patterns in chronic older patients, potentially inappropriate prescribing and adverse drug reactions: protocol of the multicentre prospective cohort study MoPIM. BMJ Open. 2020 Jan 26;10(1):e033322. doi: 10.1136/bmjopen-2019-033322. PMID 31988230
- [Derived] Ortonobes S, Herranz S, Lleal M, Sevilla-Sanchez D, Jordana R, Mascaro O, Ferrandez O, de Jaime E, Estrada R, Nazco GJ, Bare M; MoPIM Study Group. Multidisciplinary medication review during older patient hospitalization according to STOPP/START criteria reduces potentially inappropriate prescriptions: MoPIM cohort study. BMC Geriatr. 2024 Jul 8;24(1):584. doi: 10.1186/s12877-024-05185-w. PMID 38978009
- [Derived] Lleal M, Bare M, Ortonobes S, Sevilla-Sanchez D, Jordana R, Herranz S, Gorgas MQ, Espaulella-Ferrer M, Arellano M, de Antonio M, Nazco GJ, Hernandez-Luis R, On Behalf Of The MoPIM Study Group. Comprehensive Multimorbidity Patterns in Older Patients Are Associated with Quality Indicators of Medication-MoPIM Cohort Study. Int J Environ Res Public Health. 2022 Nov 29;19(23):15902. doi: 10.3390/ijerph192315902. PMID 36497976
- [Derived] Bare M, Lleal M, Ortonobes S, Gorgas MQ, Sevilla-Sanchez D, Carballo N, De Jaime E, Herranz S; MoPIM study group. Factors associated to potentially inappropriate prescribing in older patients according to STOPP/START criteria: MoPIM multicentre cohort study. BMC Geriatr. 2022 Jan 11;22(1):44. doi: 10.1186/s12877-021-02715-8. PMID 35016636
- [Derived] Bare M, Herranz S, Roso-Llorach A, Jordana R, Violan C, Lleal M, Roura-Poch P, Arellano M, Estrada R, Nazco GJ; MoPIM study group. Multimorbidity patterns of chronic conditions and geriatric syndromes in older patients from the MoPIM multicentre cohort study. BMJ Open. 2021 Nov 15;11(11):e049334. doi: 10.1136/bmjopen-2021-049334. PMID 34782339